CLINICAL TRIAL: NCT05492669
Title: Effect of Prolonging Intravenous Lidocaine on Chronic Pain and Long-term Quality of Life in Patients Undergoing Hepatectomy
Brief Title: Intravenous Lidocaine on Chronic Pain in Patients Undergoing Hepatectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-571
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Chronic Pain
Keywords: lidocaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Injections; Saline Solution

STUDY DESIGN:
Intervention Model Description: The experimental group received lidocaine and the control group received the same amount of saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants, the anesthesiologist, data collectors, the physicians performing the follow-up, and data analysts will be blinded to the group allocation. Blinding will maintain until the completion of the final analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): General anesthesia is induced in the lidocaine group with intravenous lidocaine 1.5mg/kg for ten minutes, followed by continuous injection of lidocaine 1.5mg/kg.h. At the end of the operation, the patient controlled intravenous analgesia with lidocaine is used, and the dose of lidocaine is 30mg/kg(no more than 2000mg at most).
  Interventions: Drug: Lidocaine Hydrochloride, Injectable
- Conventional analgesia group (Placebo Comparator): The lidocaine is replaced by identical volumes and rates of 0.9% saline. At the end of the operation, the patient controlled intravenous analgesia without lidocaine is used.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: Lidocaine Hydrochloride, Injectable — In the lidocaine group, at the end of the induction of general anesthesia, a bolus injection of lidocaine 1.5 mg/kg, calculated using the patient's ideal body weight and given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery. Postoperative pain management during the first 72 postoperative hours will involve the use of a PCIA device, which will contain lidocaine 30mg/kg, sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9 % normal saline.
  Other Names: lidocaine group
  Arms: Lidocaine group
Drug: 0.9% normal saline — In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2 μg/kg, granisetron 12 mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 ml.
  Other Names: placebo group
  Arms: Conventional analgesia group

SUMMARY:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT04295330 to further evaluate the effect of long-term infusion of lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing liver cancer surgery.

DETAILED DESCRIPTION:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT04295330 to further evaluate the effect of long-term infusion of lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing liver cancer surgery. 272 patients with primary liver cancer who meet the inclusion criteria are included. According to the random number, the patients are divided into lidocaine group and conventional analgesia group.In the lidocaine group, a bolus injection of lidocaine 1.5 mg/kg, given as an infusion over 10 minutes, followed by a continuous infusion of lidocaine at 1.5 mg/kg per hour for the whole surgical procedure and will be discontinued at the end of surgery. Postoperative pain management during the first 72 postoperative hours will involve the use of a PCIA device, which will contain lidocaine , sufentanil , granisetron diluted to 200 mL in 0.9 % normal saline. In the placebo group, the same volume of normal saline instead of lidocaine will be administered. Blood samples will be drawn immediately after the bolus infusion of lidocaine, at the end of surgery, and 24 hours after surgery to measure plasma lidocaine concentrations. Blood samples will also be collected at 24 hours after surgery for subsequent measurement of inflammatory factors. Numeric rating scale(NRS) is used to evaluate pain at rest and light activities at postoperative 24, 48, 72 hours. The recovery time of postoperative gastrointestinal function, length of hospital stay, and the incidence of lidocaine toxicity within postoperative 72 hours will be recorded. Follow-up after discharge includes chronic pain, the impact of chronic pain on quality of life, the relapse-free survival and overall survival from postoperative 3 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-80 years old American Society of Anesthesiologists(ASA) Ⅰ～III BMI≤30 Primary single hepatocellular carcinoma resection was proposed for patients undergoing laparotomy (median incision, right subcostal incision/inverted L-shaped incision)

Exclusion Criteria:

Primary liver cancer with malignant tumors of other organs (such as lung, kidney, intestine, etc.).

Primary hepatocellular carcinoma with portal vein or inferior vena cava and other large vascular thrombus.

Long-term opioid use, alcohol or drug abuse or any of the drugs (lidocaine, etc.) used in this study were contraindicated and allergic for patients.

Patients with severe hepatic and renal dysfunction (total bilirubin >1.46mg/dl, glomerular filtration rate <30ml/min /1.73㎡ or end-stage renal disease).

Severe heart disease (severe heart block (including sinoatrial, atrioventricular, and intraventricular block); Severe heart failure (ejection fraction <20%); Sinus bradycardia; Patients with Adams-Stokes syndrome, preexcitation syndrome, etc Patients with a history of uncontrolled seizures or acute porphyria. Long-term use of cimetidine and β-blockers (lidocaine metabolism is inhibited through the liver, resulting in increased blood concentration of the drug, which can lead to adverse cardiac and nervous system reactions).

Patients treated with drugs that are contraindicated with lidocaine (phenobarbital, thiopental, sodium nitroprusside, mannitol, amphotericin B, ampicillin, mesonotal, sulfadiazine sodium); Patients who are using enoxacin, lomefloxacin, norfloxacin, and prulifloxacin.

Patients with a history of gastrointestinal bleeding or perforation after nsaids;Patients with active gastrointestinal ulcers/bleeding or who have had recurrent ulcers/bleeding in the past.

Patients who had taken other experimental drugs or were participating or participating in other clinical trials within 3 months of enrollment.

Failure to cooperate with the study for any reason or the researcher considers it inappropriate to be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-07-27 (Estimated); Study Completion 2024-07-27 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic pain at 3 months postoperatively | 3 months postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience. The impact of chronic pain on the quality of life is also assessed by Brief Pain Inventory score.

SECONDARY OUTCOMES:
The incidence of chronic pain at 6 months ,1 year,3 year and 5 year postoperatively | 6 months, 1 year and 3 year postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience. The impact of chronic pain on the quality of life is also assessed by Brief Pain Inventory score.
The levels of inflammatory factors at 24 hours after surgery | 24 hours postoperatively
  Peripheral blood TNF-α, CXCL10, cytokines IL-6, three tumor progressions and metastasis-related markers (VEGF-A,MMP-3, MMP-9,MMP-2) etc. are measured 24 hours after operation.
The incidence of moderate to severe pain at 24, 48 and 72 hours after surgery at rest and during movement; | At 3 days after surgery
  The pain is evaluated using numerical rating scale（NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points.
The cumulative morphine consumption at 24, 48 and 72 hours postoperatively | At the end of the surgery，24，48 and 72 hours after surgery
  Intraoperative and postoperative opioid use is reported as morphine milligram equivalents, calculated using the Practical Pain Management calculator.
The incidence of a composite of postoperative pulmonary complications during | during the period from the end of surgery to discharge
  defined as positive if any component developed before discharge after surgery; These complications included respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, or aspiration pneumonitis loading dose, immediately after the end of surgery, and at the first 24 hours after surgery.
Length of hospital stay | during the period from the end of surgery to discharge
  determined by the number of days from admittance to discharge.
Plasma lidocaine concentration immediately after loading，after surgery and 24-hours postoperatively | Immediately after bolus, after surgery and 24-hour postoperatively
  Plasma lidocaine concentration is an important indicator for evaluating the safety of the drug during use.
The incidence of lidocaine toxicity within 72 hours after operation | within 72 hours after operation
  Lidocaine toxicity mainly includes neurological manifestations such as dizziness, tinnitus, convulsions, cardiac manifestations such as bradycardia, new severe atrioventricular block and so on.
Overall survival after surgery | 6 months, 1 year, 3 years, 5 years postoperatively
  Overall survival is defined as the time between the date from surgery to the date of death.
Recurrence-free survival after surgery | 6 months, 1 year, 3 years, 5 years postoperatively
  Postoperative re-examination is based on the diagnosis of enhanced CT, MRI, ultrasound or blood examination to determine whether the patient has recurrence and metastasis. Recurrence-free time refers to the time from surgery to tumor recurrence based on the above CT, MRI, etc.
Disability-free surviva survival | 6 months, 1 year, 3 years, 5 years postoperatively
  Patient self-assessment is carried out by using the World Health Organization(WHO) Disability Scale, with a minimum score of 12 points and a maximum score of 60 points. The lower the score, the higher the quality of life.

OTHER OUTCOMES:
The prevalence of neuropathic pain | 3 months, 6 months, 1 year, 3 years, 5 years postoperatively
  The ID Pain scale is used as a validated assessment of neuropathic pain. ID pain questionnaire consists of six items. Pain higher scores suggest a neuropathic component to the pain.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No